CLINICAL TRIAL: NCT02876042
Title: BAROSTIM THERAPY ™ in Heart Failure With Preserved Ejection Fraction: A Post-Market Registry With the CE-Marked BAROSTIM NEO™ System
Brief Title: BAROSTIM THERAPY™ In Heart Failure With Preserved Ejection Fraction
Acronym: HFpEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 360047-001
Record Dates: First submitted 2016-08-15; First posted 2016-08-23 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: BAROSTIM NEO™ System — Implantation of the BAROSTIM NEO™ System

SUMMARY:
The purpose of this registry (NCT02876042) is to evaluate the effect of BAROSTIM THERAPY with the BAROSTIM NEO system in the commercial setting in subjects recently implanted under the CE-Marked indication for resistant hypertension that also have evidence of heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
Summary:

The CVRx BAROSTIM THERAPY in Heart Failure with Preserved Ejection Fraction (HFpEF) Registry will be performed with subjects who have been recently implanted with the BAROSTIM NEO System in accordance with CE-Mark approved criteria for resistant hypertension and have evidence of HFpEF per the registry enrollment criteria. Subjects must be enrolled within 30 days from implant but prior to therapy activation. Up to 70 subjects will be enrolled at up to 10 sites. Data should be obtained from standard of care measurements taken prior to implant, at enrollment/baseline, and at 3 and 6 months after the device was implanted, at which time each subject will be exited from the registry.

Eligibility Criteria:

The CE-Mark approved indications and contraindications for the BAROSTIM NEO system in the treatment of resistant hypertension include:

* Indications

  * Systolic blood pressure greater than or equal to 140 mmHg, and
  * Resistance to maximally tolerated therapy with a diuretic and two other anti-hypertension medications
* Contraindications

  * Bilateral carotid bifurcations located above the level of the mandible
  * Baroreflex failure or autonomic neuropathy
  * Uncontrolled, symptomatic cardiac bradyarrhythmias
  * Carotid atherosclerosis that is determined by ultrasound or angiographic evaluation to be greater than 50%
  * Ulcerative plaques in the carotid artery as determined by ultrasound or angiographic evaluation

ELIGIBILITY:
Inclusion Criteria:

* Sign an Ethics Committee (EC) approved informed consent form for the registry.
* Implanted with the BAROSTIM NEO system in accordance with CE-Mark approved indications and contraindications for resistant hypertension within 30 days prior to enrollment.
* BAROSTIM THERAPY not yet chronically activated.
* Pre-implant echocardiogram with left ventricular ejection fraction ≥ 50% within 30 days prior to implant.
* On stable, maximally-tolerated, guideline-directed cardiovascular medications for at least 30 days prior to enrollment.
* Objective evidence of heart failure according to the following criteria:

  * Hospitalization for heart failure within 12 months prior to enrollment OR
  * Echocardiographic evidence of diastolic dysfunction (LA Volume Index >34 ml/m2 OR E/e >13) within 30 days prior to enrollment OR
  * NTproBNP > 220 pg/mL or BNP > 80 pg/mL (in atrial fibrillation, NTproBNP > 600 pg/mL or BNP > 200 pg/mL) within 30 days prior to enrollment

Exclusion Criteria:

* Heart failure secondary to a reversible or treatable condition such as, cardiac structural valvular disease, acute myocarditis and pericardial constriction.
* Heart failure secondary to right ventricular failure or right ventricular myocardial infarction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The CVRx BAROSTIM THERAPY in Heart Failure with Preserved Ejection Fraction (HFpEF) Registry will be performed with subjects who have been recently implanted with the BAROSTIM NEO System in accordance with CE-Mark approved criteria for resistant hypertension and have evidence of HFpEF per the registry enrollment criteria.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Changes in Office Cuff Systolic Blood Pressure | Pre-implant baseline to 6 months post-implant
  Office cuff blood pressure measurement to be obtained from a time point prior to implant and as close to the implant procedure as possible (baseline), and at 3 and 6 months post-implant.

SECONDARY OUTCOMES:
Change in New York Heart Association Functional Classification | Pre-implant baseline to 6 months post-implant
  New York Heart Association Classification, if available, should be obtained from a time point prior to implant and as close to the implant procedure as possible (baseline), and at 3 and 6 months post-implant.
Changes in Left Ventricular Mass Index | Pre-implant baseline to 6 months post-implant
  An echocardiogram obtained prior to implant, and as close to the implant procedure as possible, will be utilized for the baseline measurement. An additional echocardiogram will be obtained at 3 and 6 months post-implant.
Changes in LA volume index | Pre-implant baseline to 6 months post-implant
  An echocardiogram obtained prior to implant, and as close to the implant procedure as possible, will be utilized for the baseline measurement. An additional echocardiogram will be obtained at 3 and 6 months post-implant.
Changes in E/E' ratio | Pre-implant baseline to 6 months post-implant
  An echocardiogram obtained prior to implant, and as close to the implant procedure as possible, will be utilized for the baseline measurement. An additional echocardiogram will be obtained at 3 and 6 months post-implant.
Changes in NT-proBNP | Pre-implant baseline, 6 months post-implant
  If available, measurement should be obtained from a time point prior to implant and as close to the implant procedure as possible (baseline), and at 3 and 6 months post-implant.
Evaluate health care utilization over follow-up, such as heart failure hospitalizations | Pre-implant baseline to 6 months post-implant
  Health care utilization information is collected throughout follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Burkert Pieske, PhD, Study Chair — Universitätmedizin Berlin - Charité
Locations (13):
- Germany (13):
  - Berlin Charité & Deutschen Herzzentrum Berlin, Berlin
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau
  - Universitätsklinikum Köln Herzzentrum, Cologne
  - Lippe Klinikum, Detmold
  - Uniklinik Frankfurt, Frankfurt
  - Universitätsklinikum Gießen und Marburg, Giessen
  - Herzzentrum Göttingen, Göttingen
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Uniklinik Heidelberg, Heidelberg
  - Kardiologie im Klinikum Ingolstadt, Ingolstadt
  - Universitätsklinikum Regensburg, Regensburg
  - Marienkrankenhaus Siegen, Siegen

REFERENCES:
- [Background] Georgakopoulos D, Little WC, Abraham WT, Weaver FA, Zile MR. Chronic baroreflex activation: a potential therapeutic approach to heart failure with preserved ejection fraction. J Card Fail. 2011 Feb;17(2):167-78. doi: 10.1016/j.cardfail.2010.09.004. Epub 2010 Oct 29. PMID 21300307
- See also: BAROSTIM THERAPY website — https://www.barostimtherapy.com/